CLINICAL TRIAL: NCT07013422
Title: The Effectiveness of Psychoeducational Intervention in Reducing Anxiety, Depression, and Symptom Burden Among Omani Women Diagnosed With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Qaboos Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: cccrc-15-2022
Record Dates: First submitted 2025-06-01; First posted 2025-06-10 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3)
Keywords: Psychoeducational intervention; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, the Intervention Group: Received five individual psychoeducational sessions (60-90 minutes each) covering health education, stress management, coping strategies, and communication with children
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Intervention: five individual psychoeducational sessions (60-90 minutes each) coverin (Experimental): Eligible participants allocated to this arm received five individual psychoeducational sessions (60-90 minutes each) covering health education, stress management, coping strategies, and communication with children. Below is a description of the topics that were discussed with the participants in each session:
  1. First session: (Overview of treatment modalities (chemo, radiotherapy, hormonal therapy), side effects (e.g., fatigue, nausea, hair loss), and general coping strategies (e.g., diet, relaxation).
  2. second session: (Emotional preparation for mastectomy or reconstructive surgery and post-surgical care.)
  3. Third session: (Fertility, reproductive health, and strategies for managing fertility-related distress.)
  4. Fourth session: (Managing psychological impact: stress, negative thoughts, and emotional burden.)
  5. Fifth session: (Communication with children about the illness, including cultural and emotional aspects.)
  Interventions: Other: Psychoeducational support
- the Control arm: Participants Received standard medical care with no added psychoeducational content (No Intervention): the Control arm: Participants Received standard medical care with no added psychoeducational content

INTERVENTIONS:
Other: Psychoeducational support — Study Intervention: psychoeducational sessions, 5 sessions were given to the participants allocated to the intervention arm (60-90 minutes each) covering health education, stress management, coping strategies, and communication with children
  Arms: Study Intervention: five individual psychoeducational sessions (60-90 minutes each) coverin

SUMMARY:
The goal of this clinical trial is to learn if psychoeducational intervention (tailored education, coping strategies, and guided disease disclosure) in a culturally appropriate format is beneficial in Reducing Anxiety, Depression, and Symptom Burden Among Omani Women Diagnosed with Breast Cancer. Patients receiving the intervention will be compared to Women who received standard medical care with no added psychoeducational content.

DETAILED DESCRIPTION:
Eligible participants were identified through the hospital's Health Information System (HIS).

Screening was conducted by the principal researcher in collaboration with a senior oncology nurse and was based on pre-established inclusion and exclusion criteria. This included reviewing the patients' diagnosis, cancer stage, psychiatric and cognitive status, and demographic characteristics.

Patients who met the criteria were approached during their chemotherapy sessions in private treatment rooms. An information sheet was provided, the purpose of the study was explained verbally in Arabic and written informed consent was obtained. Baseline assessments (Hospital Anxiety and Depression Scale (HADS) and Edmonton Symptom Assessment Scale (ESAS)) were administered immediately after consent during the same visit.

* Structure and Content of the Intervention:

1. First session: duration 30-40 minutes Overview of treatment modalities (chemo, radiotherapy, hormonal therapy), side effects (e.g., fatigue, nausea, hair loss), and general coping strategies (e.g., diet, relaxation). 2nd session: 30-40 minutes Emotional preparation for mastectomy or reconstructive surgery and post-surgical care. 3rd session: 30-40 minutes Fertility, reproductive health, and strategies for managing fertility-related distress. 4th session : 30-40 minutes Managing psychological impact: stress, negative thoughts, and emotional burden. 5th session: 30-40 minutes Communication with children about the illness, including cultural and emotional aspects.

Delivery Technique of the Intervention:

The delivery of the psychoeducational intervention adhered to a structured yet adaptable approach, carefully aligned with the clinical routines of the daycare chemotherapy unit and the individual needs of each participant. At the beginning of each working day, the researcher accessed the hospital's Health Information System (HIS) to review the list of patients scheduled for chemotherapy. Participants in the intervention group were identified and matched against a pre-maintained tracking table documenting the session number and completion date for each participant. This system enabled the researcher to ascertain which individuals were due for a session and to plan the timing, accordingly, ensuring alignment with the patients' treatment schedules and physical conditions. Sessions were conducted individually in the private treatment rooms designated for chemotherapy administration. These rooms provided a quiet and comfortable environment conducive to privacy and uninterrupted engagement. The scheduling of each session was organized to avoid interference with medical care and to accommodate each participant's level of alertness and energy. Upon entering the room, the researcher greeted the participant with warmth and respect, briefly assessed their physical state, and began with an open-ended emotional and clinical check-in. This process involved inquiring about the participant's feelings since the last session, any emerging or worsening side effects, and whether they had reflected upon or applied any of the previously discussed topics. These follow-up conversations facilitated continuity between sessions and permitted the researcher to adapt the day's content based on the participant's current condition. The sessions were delivered verbally in Arabic, utilizing a conversational and empathetic tone. No printed handouts or written materials were provided to the participants. The researcher explained each topic using clear, accessible language, frequently pausing to check for understanding or emotional responses. Participants were encouraged to pose questions or share their thoughts, but were never pressured to engage if they preferred to remain silent.

The atmosphere was intentionally designed to be supportive, respectful, and emotionally safe.

Each session adhered to a thematic structure based on the intervention protocol, but the delivery remained flexible, contingent upon the participant's level of engagement and energy.

Some participants completed one session per week; others required longer intervals due to fatigue, low immunity, or interruptions in treatment. In certain cases, sessions were spaced up to three weeks apart. This flexibility allowed each participant to engage at her own pace without feeling overwhelmed. Subsequent to each session, the researcher documented the date, session number, approximate duration, and a brief summary of the participant's response. Observations regarding emotional readiness, questions raised, and any challenges encountered were also recorded. These records were reviewed during periodic supervision sessions with the consultant psychiatrist, who provided oversight and guidance for managing sensitive emotional content or complex patient reactions. If at any point the researcher noted that a participant was experiencing psychological distress beyond the intervention's scope-for instance, persistent sadness, anxiety, or observable signs of emotional dysregulation-the participant was promptly referred to a qualified psychiatrist or psychologist at the center for specialized support. All referrals were conducted discreetly, with full respect for the participant's privacy and comfort. This delivery technique facilitated the intervention's maintenance of both fidelity and flexibility-ensuring that core content was delivered consistently while adapting to the personal, emotional, and medical realities of each participant.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years
* Diagnosed with Stage I-III breast cancer
* Receiving chemotherapy at SQCCCRC during the study period

Exclusion Criteria:

* Non-Omani nationality
* Stage IV disease
* Major psychiatric or cognitive disorders, based on medical records

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — only biological females are eligible to participate in the study
Enrollment: 58 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-04-18 (Actual)

PRIMARY OUTCOMES:
Anxiety and depression using the Hospital Anxiety and Depression Scale (HADS) | At baseline the time of the first chemotherapy session and at 9 months follow-up
  Anxiety and depression using the Hospital Anxiety and Depression Scale (HADS) Anxiety and depression measured using the Hospital Anxiety and Depression Scale (HADS).
  Each subscale consists of 7 items scored from 0 to 3, with total scores ranging from 0 to 21. Higher scores indicate greater anxiety or depression.

SECONDARY OUTCOMES:
Symptom burden using the Edmonton Symptom Assessment Scale (ESAS) | At baseline the time of the first chemotherapy session and at 9 months follow-up
  Symptom burden using the Edmonton Symptom Assessment Scale (ESAS) Symptom burden measured using the Edmonton Symptom Assessment Scale (ESAS).
  Each symptom is rated on a scale from 0 (no symptom) to 10 (worst severity), with total scores ranging from 0 to 90. Higher scores indicate greater symptom burden.

CONTACTS AND LOCATIONS:
Locations (1):
- Sultan Qaboos Comprehensive Cancer Care and Research Centre (SQCCCRC), Muscat, Oman, Muscat, Oman